CLINICAL TRIAL: NCT00987974
Title: Short Term Statin Treatment and Endothelial Dysfunction Due to Ischemia and Reperfusion Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G. Rongen, RUNMC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMD01
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2001-04

CONDITIONS: Ischemia Reperfusion Injury; Endothelial Dysfunction
Keywords: ischemia reperfusion injury; endothelial dysfunction; statins; rosuvastatin; atorvastatin; placebo; ecto-5'-nucleotidase; flow mediated dilation
MeSH Terms: conditions — Reperfusion Injury | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- rosuvastatin 3days (Experimental): 8 Subjects will use rosuvastatin 20 mg/day for 3 days
  Interventions: Drug: rosuvastatin
- atorvastatin 3 days (Active Comparator): 8 Subjects will use atorvastatin 80 mg/day for 3 days.pj
  Interventions: Drug: atorvastatin 3 days
- placebo 3days (Placebo Comparator): 8 Subjects will use placebo for 3 days.
  Interventions: Drug: placebo
- rosuvastatin 7 days (Experimental): 8 Subjects will use rosuvastatin 20 mg/day for 7 days.
  Interventions: Drug: rosuvastatin 7 days
- atorvastatin 7 days (Active Comparator): 8 Subjects will use atorvastatin 80 mg/day for 7 days.
  Interventions: Drug: atorvastatin 7 days
- placebo 7 days (Placebo Comparator): 8 Subjects will use placebo for 7 days.
  Interventions: Drug: placebo 7 days

INTERVENTIONS:
Drug: rosuvastatin — rosuvastatin 20 mg/day for 3 days.
  Other Names: crestor
  Arms: rosuvastatin 3days
Drug: atorvastatin 3 days — atorvastatin 80 mg/day for 3 days.
  Other Names: lipitor
  Arms: atorvastatin 3 days
Drug: placebo — placebo for 3 days.
  Arms: placebo 3days
Drug: rosuvastatin 7 days — rosuvastatin 20 mg/day for 7 days
  Other Names: crestor
  Arms: rosuvastatin 7 days
Drug: atorvastatin 7 days — atorvastatin 80 mg/day for 7 days.
  Other Names: lipitor
  Arms: atorvastatin 7 days
Drug: placebo 7 days — placebo 7 days
  Arms: placebo 7 days

SUMMARY:
Rationale:

Apart from their cholesterol lowering effects, statins have cholesterol-independent pleiotropic actions, such as upregulation of 5'-ectonucleotidase and up-regulation of NO-synthase that may increase tolerance against ischemia-reperfusion injury (IR-injury). Several animal studies have shown reduction of IR-injury as a result of statin treatment in both the heart and the kidney. Recently the investigators have shown, using Annexin A5 targeting after voluntary ischemic exercise to assess IR-injury, a protective effect of a 7 day oral rosuvastatin treatment. A three day treatment with atorvastatin however failed to reduce annexin targeting.

Assessment of the flow mediated dilation of the brachial artery as measure of endothelial (dys)function, is a validated model to research effects of possible protective strategies and perform mechanistic experiments on IR-injury in humans in vivo.

The investigators hypothesize that pretreatment with statins can increase endothelial tolerance against ischemia and reperfusion injury.

Objective:

To study the protective effect of pretreatment (both 3 day and 7 day) with rosuvastatin and atorvastatin on flow mediated dilation after 15 minutes ischemia and 15 minutes reperfusion.

Study design: placebo-controlled randomised double-blind trial

Study population: Healthy volunteers, age 18-50

Intervention: Treatment with either rosuvastatin 20 mg, atorvastatin 80mg or placebo during either 3 or 7 days

Main study parameters: Difference in flow mediated dilation before and after 15 minutes ischemia.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Treatment with rosuvastatin or atorvastatin is not expected to harm the volunteers. Most reported side effects of rosuvastatin and atorvastatin are gastro-intestinal complains and myalgia. The volunteers will not benefit directly from participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Written informed consent

Exclusion Criteria:

* Smoking
* History of any cardiovascular disease
* Hypertension (in supine position: systole >140 mmHg, diastole >90 mmHg)
* Diabetes Mellitus (fasting glucose >7.0 mmol/L or random glucose >11.0 mmol/L)
* Hyperlipidaemia (fasting total cholesterol >5.5 mmol/L or random cholesterol >6.5 mmol/L)
* Alanine amino transferase >90 U/L
* Creatine kinase >440 U/L
* Raised rhabdomyolysis risk

  * GFR <60 ml/min
  * Overt clinical signs of hypothyroidism
  * Myopathy in family history
  * Alcohol abuse
* Concomitant chronic use of medication
* Participation to any drug-investigation during the previous 60 days as checked with VIP check.
* Professional athletes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Difference in flow mediated dilation before and after 15 minutes ischemia | 30 minutes

SECONDARY OUTCOMES:
Ecto-5'-nucleotidase activity and lipid profile after statin therapy | 3-7 days

CONTACTS AND LOCATIONS:
Locations (1):
- RUNMC, Nijmegen, Netherlands

REFERENCES:
- [Background] Meijer P, Oyen WJ, Dekker D, van den Broek PH, Wouters CW, Boerman OC, Scheffer GJ, Smits P, Rongen GA. Rosuvastatin increases extracellular adenosine formation in humans in vivo: a new perspective on cardiovascular protection. Arterioscler Thromb Vasc Biol. 2009 Jun;29(6):963-8. doi: 10.1161/ATVBAHA.108.179622. Epub 2009 Apr 9. PMID 19359665
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Derived] Wouters CW, Wever KE, Bronckers I, Hopman MT, Smits P, Thijssen DH, Rongen GA. Short-term statin treatment does not prevent ischemia and reperfusion-induced endothelial dysfunction in humans. J Cardiovasc Pharmacol. 2012 Jan;59(1):22-8. doi: 10.1097/FJC.0b013e318232b1a4. PMID 21885990